CLINICAL TRIAL: NCT03926078
Title: Three-dimensional Optical Surface Imaging as a Diagnostic Tool for Severity Quantification and Clinical Decision Making in Pectus Excavatum
Brief Title: Three-dimensional Optical Surface Imaging as a Diagnostic Tool in Pectus Excavatum
Acronym: 3D PECTUS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Zuyderland Medisch Centrum (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: Single | Purpose: Diagnostic
Other Study IDs: METCZ20190048
Record Dates: First submitted 2019-04-18; First posted 2019-04-24 (Actual); Last update posted 2020-07-02 (Actual); Status verified 2020-07

CONDITIONS: Pectus Excavatum
Keywords: Haller Index; Optical Imaging; Torso Topography; Three-dimensional Surface Scan; Diagnostic accuracy
MeSH Terms: conditions — Funnel Chest | interventions — X-Rays

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: All measurements will be performed by three blinded observers that are not responsible to perform a comprehensive interpretation of the study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Patients under 18 years of age (Other): Group A consists of patients that receive a chest radiography in the current work-up of PE.
  Interventions: Other: 3D optical surface image; Radiation: Chest radiography
- Patients aged 18 years or older (Other): Group B consists of patients that receive a CT scan in the current work-up of PE.
  Interventions: Other: 3D optical surface image; Radiation: CT scan

INTERVENTIONS:
Other: 3D optical surface image — 3D optical surface images will be acquired and used to calculate the EHI
Radiation: Chest radiography — Chest radiographies will be acquired and used to calculated the HI and EHI
  Arms: Patients under 18 years of age
Radiation: CT scan — CT scans will be acquired and used to calculate the HI and EHI
  Arms: Patients aged 18 years or older

SUMMARY:
Pectus excavatum (PE) is the most common anterior chest wall deformity. Currently, a chest radiography (CR) or Computed Tomography (CT) scan is acquired to determine and objectify pectus severity using the Haller Index. Alongside other determinants, the Haller Index value is used in the proces of clinical decision making and determine surgical candidacy. However, cross-sectional imaging based calculation of the Haller Index implies exposure to ionizing radiation that should be limited at all times to diminish the cumulative long-term risks of malignancy. Especially in pectus patients that often concerns children.

Three-dimensional (3D) optical surface imaging offers a non-invasive, radiation-free alternative that may be used to obtain thoracic measures and determine pectus severity. However, for 3D images/scans to be used as a diagnostic tool in the proces of clinical decision making and determine surgical candidacy, its diagnostic accuracy should be evaluated. This will be investigated utilizing a pilot study design as no prior accuracy studies are available.

DETAILED DESCRIPTION:
This single-centre prospective pilot study is conducted to assess the diagnostic accuracy of 3D optical surface imaging based external Haller Index (EHI) measurements to quantify the severity of pectus excavatum. CR and CT based conventional Haller Indices (HI) are used as reference method.

CR and CT are both used as reference method, as the work-up of pectus patients in our centre is dependent of age. Subsequently, two groups are created: (A) patients under 18 years of age that receive a frontal (anteroposterior) and sagittal chest radiography, and (B) patients aged 18 years or older that receive a chest CT scan.

In this study, patients are their own control. To obtain optical surface images, a handheld 3D scanner is used. During acquisition, subjects will be standing in an upright position with arms abducted. Standard routinely used protocols are used to acquire chest radiographies and CT scans.

The HI is obtained from all chest radiographies and CT scans, calculated by dividing the widest thoracic transverse diameter by the anteroposterior distance, measured from the posterior surface of sternum to the anterior surface of the vertebral body. The EHI, a modified measurement to assess pectus deformity, is used to quantify PE severity based on 3D optical surface images. The EHI is calculated by dividing the widest external thoracic transverse diameter by the distance between the external deepest point or point of maximal protrusion and external vertebral body. The EHI is also calculated from the available chest radiographies and CT scans.

All measurements will be performed by three blinded observers that are not responsible to perform a comprehensive interpretation of the study. Following acquisition of all indices, the inter-observer reliability is calculated using the intraclass correlation coefficient. Based on the means, a receiver-operating characteristic (ROC)-curve is created for the 3D scan based EHI measurements, utilizing the surgical indication based on CR and CT (HI larger or equal to 3.25) images as gold standard. The optimal cut-off value, obtained from the ROC-curve is subsequently used to determine the 3D optical surface images' diagnostic accuracy.

ELIGIBILITY:
Inclusion criteria:

* All patients that visit the Zuyderland Medical Centre outpatient clinic for evaluation of their pectus excavatum.
* No age restrictions were imposed, however, to be eligible, it was mandatory to be able to stand still in and upright position for 60 seconds.

Exclusion criteria:

- Patients that suffer from any form of light hypersensitivity or epilepsy were not considered while 3D optical surface images were acquired with the use of structured, flashing light.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 28 (Estimated)
Dates: Start 2019-08-21 (Actual); Primary Completion 2021-02 (Estimated); Study Completion 2021-03 (Estimated)

PRIMARY OUTCOMES:
Diagnostic accuracy of the EHI, calculated from 3D optical surface images | 1 year
  Dependent of age, the CR or CT based HI is utilized as reference method

SECONDARY OUTCOMES:
Inter-observer reliability | 1 year
  Inter-observer reliability of CR, CT and 3D image derived (external) Haller Inidices, obtained by 3 observers
Correlation of CT scan derived HI and EHI | 1 year
  Correlation is assessed by the Pearson's correlation coefficient
Correlation of CT scan derived EHI and 3D optical surface image derived EHI | 1 year
  Correlation is assessed by the Pearson's correlation coefficient
Correlation of CT and CR derived HI with 3D optical surface image derived EHI | 1 year
  Correlation is assessed by the Pearson's correlation coefficient
Absolute agreement of CT scan derived EHI and 3D optical surface image derived EHI | 1 year
  Assessed by the intraclass correlation coefficient

CONTACTS AND LOCATIONS:
Locations (1):
- Zuyderland Medical Centre, Heerlen, Limburg, Netherlands